CLINICAL TRIAL: NCT06901336
Title: An Open-Label Phase 1 Study in Healthy Male Subjects to Investigate the Absorption, Distribution, Metabolism and Excretion of [14C]-STX-478 Following Single-Dose Oral Administration
Brief Title: A Study of LY4064809 [14C]-STX-478 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scorpion Therapeutics, a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 27692; J6M-MC-JSGB (Other: Eli Lilly and Company); STX-478-102 (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-03-24; First posted 2025-03-28 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-STX-478 (Experimental): Healthy participants will receive a single dose of [14C]-STX-478.
  Interventions: Drug: [14C]-STX-478

INTERVENTIONS:
Drug: [14C]-STX-478 — oral administration
  Other Names: LY4064809

SUMMARY:
The main purpose of this study is to conduct blood tests to measure how much STX-478 is in the bloodstream and how the body handles and eliminates it in healthy participants. This study will involve a single dose of 14C radiolabeled STX-478. This means that a radioactive tracer substance, C14, will be incorporated into the study drug STX-478 to investigate the study drug and its breakdown products and to find out how much of these passes from blood into urine, feces and expired air. The study will also evaluate the safety and tolerability of STX-478.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 18.0 kg/m2 and ≤ 32.0 kg/m2 at Screening; body weight

  ≥ 55.0 kg and ≤ 100.0 kg at Screening.
* Negative serology results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) and human immunodeficiency virus antibody and antigen (HIV Ab/Ag).
* Non-smoker (with no use of other tobacco or nicotine containing products, in any form), as documented by history (no nicotine within 6 months prior to Screening) and a negative cotinine test at Screening and admission

Exclusion Criteria:

History or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor

* Any history of serious allergic/hypersensitivity reactions
* History or presence of alcohol or drug abuse (self-reported) within 2 years prior to Screening.
* Administration of any prescription or non-prescription drugs (including antacids; however, acetaminophen at a dose ≤ 1 g/day is permitted), herbal remedies or vitamin supplements from 28 days, or five half-lives, whichever is longer, prior to Admission.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants with female sexual partner(s) of reproductive potential may be enrolled if the male:
  * is documented to be surgically sterile (i.e., successfully vasectomized) at least 90 days prior to screening; or
  * agrees to use effective contraception, for at least 90 days after receiving study drug and agrees to refrain from sperm donation from the time of Screening through 90 days post dose.
Enrollment: 8 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Percentage of the Total Radioactive Dose in Urinary, Fecal, and Urinary and Fecal Combined Excretion | Baseline, Up to Day 29

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of 14C and STX-478 | Predose up to Day 29 Post Dose
PK: Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC 0- inf) of 14C and STX-478 | Predose up to Day 29 Post Dose
Total Radioactivity Recovered in Urine and Feces | Predose up to Day 29 Post Dose
Total Number of Metabolites and Identification of Metabolites of STX-478 in Plasma, Urine, and Feces | Predose up to Day 29 Post Dose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Pharmaron Clinical Pharmacology Center Inc, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No